CLINICAL TRIAL: NCT07308951
Title: Clinical Efficacy Evaluation of Patient-Controlled Transcutaneous Electrical Acupoint Stimulation in Improving the Quality of Life for Patients With Chronic Cancer Pain
Brief Title: Effect of Patient-Controlled Transcutaneous Electrical Acupoint Stimulation on Quality of Life in Chronic Cancer Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Yi Liang, Director, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20231208064031886
Record Dates: First submitted 2025-11-29; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Quality of Life; Chronic Cancer Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS Intervention Group (Experimental): First, acupoint group ① (bilateral Hegu [LI4] and Neiguan [PC6]) received 30 minutes of transcutaneous electrical acupoint stimulation (TEAS), followed by acupoint group ② (bilateral Sanyinjiao [SP6] and Zusanli [ST36]) for the same duration.
  Interventions: Other: TEAS
- Sham TEAS Control Group (Placebo Comparator): Except for the transcutaneous acupoint electrical stimulator, which has no current output, the other operations are the same as TEAS Intervention Group.
  Interventions: Other: sham TEAS

INTERVENTIONS:
Other: TEAS — Patients assumed a supine or sitting position, and after routine skin disinfection at the acupoint sites, one pair of electrode patches was attached to the two ipsilateral acupoints of the same group, with the same procedure performed on the contralateral side. A transcutaneous electrical acupoint stimulator was used to apply TEAS sequentially to acupoint groups ① and ②. Each acupoint group received a single TEAS session lasting 30 minutes. Participants were permitted to undergo multiple TEAS sessions within the same day, with all treatments recorded in a pain diary.
  The TEAS parameters were set as a continuous wave at a frequency of 2 Hz, with the current intensity adjusted to the patient's tolerance level. The treatment followed a "patient-controlled, as-needed" administration pattern. Each treatment course lasted 7 days, with a minimum of 3 treatment days per course and a total of no fewer than 5 sessions per course. A total of 4 treatment courses were conducted.
  Arms: TEAS Intervention Group
Other: sham TEAS — Participants were informed that, due to individual variations in sensory thresholds, it is normal if no distinct sensation is perceived even at the maximum stimulation intensity. Regardless of subjective perception, the transcutaneous electrical acupoint stimulation treatment remains active and exerts its therapeutic effects continuously.
  Arms: Sham TEAS Control Group

SUMMARY:
This study aims to objectively evaluate the effect of Patient-Controlled Transcutaneous Electrical Acupoint Stimulation (PC-TEAS) on improving the quality of life in patients with chronic cancer pain, thereby providing evidence-based medical support for its efficacy and offering practical basis for patients to achieve home-based auxiliary treatment based on their own needs. Furthermore, by observing and comparing changes in indicators such as pain-related scores, analgesic consumption, emotional scores, spontaneous bowel movements, and adverse events, this research will comprehensively assess the advantages of PC-TEAS in the management of chronic cancer pain and explore other potential benefits of this intervention for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years, regardless of gender;
* Diagnosis of primary or metastatic malignant tumor confirmed by histopathology and/or cytology, consistent with the American Cancer Society criteria for malignancy;
* Presence of cancer-related pain, defined as an average Numeric Rating Scale (NRS) score ≥ 2 over the preceding week or current regular use of opioid analgesics;
* Life expectancy ≥ 3 months;
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score ≤ 2, stable vital signs, clear consciousness, intact pain perception, unimpaired communication, ability to cooperate with study procedures and complete assessments;
* Provision of signed informed consent by the patient or their legal guardian after comprehensive explanation of the study;

Exclusion Criteria:

* Pain not attributable to cancer;
* Severe cardiopulmonary dysfunction or respiratory depression;
* Implantation of cardiac pacemaker or metallic implants at stimulation sites;
* Local skin lesions or conditions unsuitable for TEAS at the acupoint sites;
* Severe psychiatric disorders or significant cognitive impairment;
* Concurrent participation in other clinical trials that may interfere with the outcome evaluation of this study;
* Previous history of transcutaneous electrical acupoint stimulation (TEAS) or transcutaneous electrical nerve stimulation (TENS);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The area under the curve (AUC) of the FACT-G (Functional Assessment of Cancer Therapy - General) total score for assessing quality of life in patients with chronic cancer pain after 4 weeks of treatment. | Baseline; Week 1; Week 2; Week 3;Week 4; Week 8; Week 12
  the FACT-G comprises 27 items grouped into 4 domains: physical well-being, social/family well-being, emotional well-being, and functional well-being; some items require reverse scoring, with the total score ranging from 0 to 108. Higher scores indicate better quality of life. Using the area under the curve scoring method allows for the observation of the cumulative benefit of PC-TEAS usage in patients over the entire treatment period

SECONDARY OUTCOMES:
the changes in BPI score from baesline | Baseline; Week 4; Week 8; Week 12
  The Brief Pain Inventory (BPI) is primarily used to assess pain severity and its multidimensional impact on patients' quality of life. The scale consists of two core components: BPI-S (Pain Severity) and BPI-I (Pain Interference). The BPI-S quantifies the severity of pain through four items: average pain, worst pain, least pain, and current pain intensity. The BPI-I evaluates the degree to which pain interferes with daily functioning across seven domains: mobility, activities of daily living, work, sleep, relationships with others, enjoyment of life, and mood, thereby providing a comprehensive multidimensional reflection of pain's impact on patient quality of life.Scores range from 0-10, with higher scores indicating more severe pain
Dosage of analgesics used on the assessment days | Baseline; Week 4; Week 8 ; Week 12
  Changes in the amount of analgesic use from baseline
Spontaneous bowel movements (SBM) during assessment days | Baseline; Week 4; Week 8; Week 12
  Spontaneous bowel movements (SBM) refer to bowel movements that occurred in the past 24 hours without the use of rescue laxatives. The number of spontaneous bowel movements by the subjects in the past week was recorded.
Bowel Function Index (BFI) during assessment days | Baseline; Week 4; Week 8; Week 12
  The Bowel Function Index (BFI) is a clinical tool specifically designed to assess opioid-induced constipation. It records the patient's ratings over the past week for straining during defecation, sense of incomplete bowel evacuation, and overall satisfaction with the bowel movement process.
The changes in mood scale scores of Hamilton Depression Rating Scale (HAMD) on the assessment days | Baseline; Week 4; Week 8;Week 12
  The Hamilton Depression Rating Scale (HAMD) is used to assess depressive. The HAMD serves as a standard clinical instrument for evaluating depressive states, In this study, participants' HAMD-17 total scores were recorded to observe changes from baseline.
The changes in mood scale scores of Hamilton Anxiety Scale (HAMA) on the assessment days | Baseline; Week 4; Week 8; Week 12
  The Hamilton Anxiety Scale (HAMA) is used to assess anxiety symptoms, The HAMA provides an important basis for diagnosing anxiety disorders and grading their severity. In this study, participants' HAMA scores were recorded to observe changes from baseline.
Frequency of breakthrough pain in the week preceding the assessment days | Baseline; Week 4;Week 8; Week 12
  The frequency of breakthrough pain episodes, along with the types and doses of rescue medication used in the preceding week, were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medicinal University, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No